CLINICAL TRIAL: NCT02260648
Title: A Double-Blind Efficacy and Safety Study of Evacetrapib in Combination With Atorvastatin in Japanese Patients With Primary Hypercholesterolemia
Brief Title: A Study of Evacetrapib (LY2484595) in Combination With Atorvastatin in Japanese Participants With Primary Hypercholesterolemia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study termination due to insufficient efficacy.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14501; I1V-JE-EIBG (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — evacetrapib; Ezetimibe; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Evacetrapib (Experimental): 130 milligrams (mg) evacetrapib and 10 mg atorvastatin administered PO once a day for 12 weeks.
  Interventions: Drug: Evacetrapib; Drug: Atorvastatin
- Ezetimibe (Active Comparator): 10 mg ezetimibe and 10 mg atorvastatin administered PO once a day for 12 weeks as a reference arm.
  Interventions: Drug: Ezetimibe; Drug: Atorvastatin
- Placebo (Placebo Comparator): Placebo and 10 mg atorvastatin administered PO once a day for 12 weeks.
  Interventions: Drug: Atorvastatin; Drug: Placebo

INTERVENTIONS:
Drug: Evacetrapib — Administered orally
  Other Names: LY2484595
  Arms: Evacetrapib
Drug: Ezetimibe — Administered orally
  Arms: Ezetimibe
Drug: Atorvastatin — Administered orally
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of the study drug known as evacetrapib when administered in combination with atorvastatin for 12 weeks in Japanese participants with primary hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* Must be treated with atorvastatin 10 mg/day for at least 30 days prior to study initiation.
* Japanese outpatients who are diagnosed with primary hypercholesterolemia with LDL-C levels (measured by a direct method) that meet the following criteria. (Participant categories are based on the definition in Japan Atherosclerosis Society 2012 guidelines.)

  * Category I: 160 mg/deciliter (dL)≤LDL-C
  * Category II: 140 mg/dL≤LDL-C
  * Category III: 120 mg/dL≤LDL-C
  * Secondary prevention: 100 mg/dL≤LDL-C
* Have triglycerides (TG) ≤400 mg/dL.
* Have HDL-C <100 mg/dL.

Exclusion Criteria:

* Participants on LDL apheresis or plasma apheresis.
* Participants with secondary hypercholesterolemia or homozygous familial hypercholesterolemia.
* Any planned angiography. If angiography is planned, participants may be screened and enrolled after all such planned procedures are completed.
* History of any of the following conditions < 90 days prior to study initiation

  * acute coronary syndrome (unstable angina, acute myocardial infarction)
  * symptomatic peripheral arterial disease
  * invasive treatment of carotid artery disease
  * ischemic stroke or transient ischemic attack (TIA)
  * intracranial hemorrhage
* History of abdominal aortic aneurysm.
* Participants with a history of intolerance/hypersensitivity to ezetimibe or statins.
* Have systolic blood pressure (SBP) > 160 millimeters of mercury (mm Hg) or diastolic blood pressure (DBP) > 100 mm Hg.
* Have a hemoglobin A1c ≥8.4% (National Glycohemoglobin Standardization Program).
* During the study period, participants who plan to use, are likely to require, or unwilling or unable to stop with adequate washout any prescription, over the counter (OTC) medication, supplements or health foods with the intent to treat serum lipids (LDL-C, HDL-C, TG) including but not limited to these classes of drugs: statin (except for atorvastatin 10 mg), ezetimibe, bile acid sequestrant, eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA). Participants taking probucol, fibrate or nicotinic agents within 8 weeks before study initiation are excluded from the study.
* Have been exposed to cholesteryl ester transfer protein (CETP) inhibitors (for example, anacetrapib or dalcetrapib).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- Japan (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ibaraki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shizuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- Evacetrapib: 130 milligram (mg) evacetrapib and 10 mg atorvastatin administered PO once a day for 12 weeks.
- Placebo: Placebo and 10 mg atorvastatin administered orally (PO) once a day for 12 weeks.
Period: Overall Study
Arm/Group | Evacetrapib | Placebo | Ezetimibe
Started | 53 | 46 | 50
Received at Least One Dose of Study Drug | 53 | 46 | 50
Completed | 35 | 33 | 42
Not Completed | 18 | 13 | 8
Not completed — Adverse Event | 3 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Discontinue Due to Study Termination | 13 | 12 | 7

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Evacetrapib: 130 mg evacetrapib and 10 mg atorvastatin administered PO once a day for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Evacetrapib | Placebo | Ezetimibe | Total
Number analyzed (Participants) | 53 | 46 | 50 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (11.53) | 57.9 (10.81) | 58.0 (10.40) | 58.2 (10.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 24 | 67
  Male | 32 | 24 | 26 | 82
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 53 | 46 | 50 | 149
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 53 | 46 | 50 | 149

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Week 12 in Low-Density Lipoprotein Cholesterol (LDL-C) Measured by Beta Quantification
Description: The mixed-effects model for repeated measures (MMRM) was used for the Least Squares Mean (LS Mean) estimates at Week 12 for LDL-C adjusting for baseline as response variables, baseline measurement as a covariate, treatment, Visit (4,5,6, or 7), and treatment-by-visit interaction as fixed effects, and participant as a random effect.
Time Frame: Baseline, Week 12
Population: All participants who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: percent change in LDL-C
Arm/Group | Evacetrapib | Placebo | Ezetimibe
Number analyzed (Participants) | 53 | 46 | 50
percent change in LDL-C | -26.37 (3.108) | -3.75 (3.264) | -27.31 (3.128)

2. Secondary Outcome: Percent Change From Baseline to Week 12 in High-Density Lipoprotein Cholesterol (HDL-C)
Description: The MMRM was used for the LS Mean estimates at Week 12 for HDL-C adjusting for baseline as response variables, baseline measurement as a covariate, treatment, visit, and treatment-by-visit interaction as fixed effects, and participant as a random effect, and treatment-by-visit interaction as fixed effects, and participant as a random effect.
Time Frame: Baseline, Week 12
Population: All participants who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: percent change in HDL-C
Arm/Group | Evacetrapib | Placebo | Ezetimibe
Number analyzed (Participants) | 53 | 46 | 50
percent change in HDL-C | 108.96 (5.150) | -0.90 (5.363) | -3.12 (5.166)

3. Secondary Outcome: Percent Change From Baseline to Week 12 in LDL-C (Direct)
Description: The MMRM was used for the LS Mean estimates at Week 12 for LDL-C (direct) adjusting for baseline as response variables, baseline measurement as a covariate, treatment, visit, and treatment-by-visit interaction as fixed effects, and participant as a random effect.
Time Frame: Baseline, Week 12
Population: All participants who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: percent change in LDL-C (Direct)
Arm/Group | Evacetrapib | Placebo | Ezetimibe
Number analyzed (Participants) | 53 | 46 | 50
percent change in LDL-C (Direct) | -27.17 (2.708) | -3.40 (2.845) | -28.96 (2.726)

4. Secondary Outcome: Percent Change From Baseline to Week 12 in Non HDL-C
Description: The MMRM was used for the LS Mean estimates at Week 12 for Non HDL-C adjusting for baseline as response variables, baseline measurement as a covariate, treatment, visit, and treatment-by-visit interaction as fixed effects, and participant as a random effect.
Time Frame: Baseline, Week 12
Population: All participants who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: percent change in non HDL-C
Arm/Group | Evacetrapib | Placebo | Ezetimibe
Number analyzed (Participants) | 53 | 46 | 50
percent change in non HDL-C | -22.01 (2.455) | -6.42 (2.577) | -27.35 (2.468)

5. Secondary Outcome: Percent Change From Baseline to Week 12 in Lipoprotein-a
Description: The analysis of covariance (ANCOVA) model using last observation carried forward (LOCF) was applied to analyze percent changes from baseline.
Time Frame: Baseline, Week 12
Population: All participants who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: percent change in Lipoprotein-a
Arm/Group | Evacetrapib | Placebo | Ezetimibe
Number analyzed (Participants) | 53 | 46 | 50
percent change in Lipoprotein-a | -33.17 (4.024) | 7.78 (3.895) | 0.68 (3.704)

6. Secondary Outcome: Percent Change From Baseline to Week 12 in Apolipoprotein A-I
Description: The ANCOVA model using last observation carried forward (LOCF) was applied to analyze percent changes from baseline.
Time Frame: Baseline, Week 12
Population: All participants who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: percent change in Apolipoprotein A-I
Arm/Group | Evacetrapib | Placebo | Ezetimibe
Number analyzed (Participants) | 53 | 46 | 50
percent change in Apolipoprotein A-I | 42.8 (2.27) | 0.6 (2.44) | -0.6 (2.34)

7. Secondary Outcome: Percent Change From Baseline to Week 12 in Apolipoprotein B
Description: The ANCOVA model using last observation carried forward (LOCF) was applied to analyze percent changes from baseline.
Time Frame: Baseline, Week 12
Population: All participants who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: percent change in Apolipoprotien B
Arm/Group | Evacetrapib | Placebo | Ezetimibe
Number analyzed (Participants) | 53 | 46 | 50
percent change in Apolipoprotien B | -20.4 (2.42) | -3.0 (2.60) | -20.4 (2.48)

ADVERSE EVENTS:
Arm/Group | Evacetrapib | Placebo | Ezetimibe
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/46 | 0/50
Other Adverse Events (participants affected / at risk) | 18/53 | 13/46 | 12/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Evacetrapib (N=53) | Placebo (N=46) | Ezetimibe (N=50)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Presbyacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Genital herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 2 (2) | 2 (2)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urethritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Mental fatigue (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema ab igne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated prematurely due to insufficient efficacy of the I1V-MC-EIAN (NCT01687998) study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days